CLINICAL TRIAL: NCT06504641
Title: Acceptability, Feasibility, and Potential Effectiveness of Video-based Patient Records for Supporting Care Delivery for Older People With Frailty.
Brief Title: I4F: Isla for Frailty Feasibility Study
Acronym: I4F
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Health Education England, Wessex (Other)
Responsible Party: Sponsor
Other Study IDs: 23SM8192
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Frailty
Keywords: Frailty; Communication; Patient assessment; Video-recording; Care transitions; Care continuity
MeSH Terms: conditions — Frailty; Communication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (3):
- Patients: Up to 30 adults, aged 65 years or older, who are frail or pre-frail, and who are admitted as an inpatient to an acute Medicine for the Elderly ward during a three-month pilot phase
  Intervention: Isla for Frailty - video-based patient records. Isla is a technology company providing a visual patient record platform. The platform allows anyone involved in a patient's care to capture and review visual data (photographs, videos) relating to a patient's health. The platform is web-based (a "progressive web application") and supports secure capture of visual data with encrypted storage in the cloud. Isla interfaces with Electronic Health Record (EHR) systems including Cerner, enabling health professionals to view data held on Isla's servers from within the electronic patient record, via the 'Cerner Red Button'. Health professionals can also view a patient's visual record through a secure weblink requiring an NHS email address and password.
  Interventions: Other: Isla for Frailty
- Carers: Carers of enrolled patients, who are in receipt of the Isla for Frailty intervention (described above)
  Carers are those who provide the enrolled patient with assistance in their daily activities and are unpaid for these caring activities. A carer may be a member of the patient's family, a friend, or other person who provides the patient with unpaid care.
  Interventions: Other: Isla for Frailty
- Ward team: Clinical staff working on one of three Medicine for the Elderly wards at St Mary's Hospital, where the Isla for Frailty intervention (described above) will be subject to a feasibility trial.
  Clinical staff must work regular shifts on the ward during study initiation and pilot phases.
  Interventions: Other: Isla for Frailty

INTERVENTIONS:
Other: Isla for Frailty — Isla for Frailty - video-based patient records. Isla is a technology company providing a visual patient record platform. The platform allows anyone involved in a patient's care to capture and review visual data (photographs, videos) relating to a patient's health. The platform is web-based (a "progressive web application") and supports secure capture of visual data with encrypted storage in the cloud.
  Isla interfaces with Electronic Health Record (EHR) systems including Cerner, enabling health professionals to view data held on Isla's servers from within the electronic patient record, via the 'Cerner Red Button'. Health professionals can also view a patient's visual record through a secure weblink requiring an NHS email address and password.

SUMMARY:
BACKGROUND: Older patients with frailty have complex support needs. How they manage with daily tasks such as eating and drinking, mobilising, communicating their preferences, and the level of support they need, can vary on a day-to-day basis. They are at risk of rapid loss of functional independence when they are acutely unwell. When older people need input from multiple different professionals, ineffective communication is sadly very common. This leads to disjointed care, and patients becoming frailer and suffering avoidable health complications. One of the problems is that it can be difficult for healthcare professionals to build up a complete picture of a patient from brief verbal handovers and written information in medical records. It is believed that video-recordings capturing the changing functional abilities and support needs of individual patients could improve care-provider communication and support for older people. Smartphones with cameras are now a part of everyday life, and people often tell their stories using photographs and videos. However, video recording patients during care delivery is not commonplace. It is not know how patients and carers feel about being video recorded or whether video recordings improve care.

AIM: To explore the perspectives of frail older patients, carers, and clinical staff around video recording during routine clinical care, and to understand how patient videos could impact on communication and care delivery across care transitions.

METHODS: The study team will recruit frail, older inpatients, their carers, and clinical staff from a Medicine for the Elderly ward. Over three months, doctors, nurses, and therapists will securely record and view patient videos alongside providing usual care. Videos will capture patients' functional abilities and support needs to inform ongoing assessment and care delivery. The investigators will collect information from patients/ carers/ doctors/ nurses /therapists about their experiences of the video recording intervention through interviews and questionnaires.

DETAILED DESCRIPTION:
Around 10% of people aged over 65 years have frailty, rising to nearly 50% of those aged over 85 years, and frailty prevalence is expected to increase alongside the growth of the ageing population.

Older people with frailty commonly require input from multiple professionals across primary, secondary, and social care. Professional bodies including the British Geriatrics Society have advocated for responsible information sharing to ensure that older people with frailty are supported to age well. Yet, as patients move between different parts of the health and care service, communication between different professionals and different providers is frequently ineffective, assessments are duplicated, and carers are repeatedly asked to provide the same information. Poorly coordinated care is linked to avoidable complications, accelerated deconditioning, and loss of independence, as well as greater carer burden and increased costs to health and social care.

Much communication across professional and organisational boundaries takes place through written referrals and (increasingly) through shared electronic patient records. Electronic health records (EHRs) are voluminous, containing large quantities of unstructured text. This plethora of data, combined with variability in documentation practices and the propagation of erroneous information in the record, means clinicians face significant challenges retrieving information to support clinical assessment. Excessive time spent in the EHR system is known to be a major source of clinician dissatisfaction contributing to stress and burnout, but failure to retrieve relevant information can lead to medical errors and poor quality care. Moreover, while text is appropriate for communicating certain types of clinical information (for example, diagnoses, comorbidities, prescribed medications, allergies, etc), it is difficult to discern the nuances of a frail older patient's condition in relation to aspects such as functional ability, cognition, behavioural symptoms, and support needs from text narratives alone. Receiving professionals may be left wondering 'Is this normal for this patient?' It is vital that health and care professionals can recognise and track subtle changes to proactively manage avoidable deconditioning and deliver individualised, person-centred care. More sophisticated modes of documentation and communication are needed to improve patient assessment and care continuity across transitions of care.

In an age of smartphones, people are increasingly telling their stories using photographs and video recordings.Technological advances allow for a variety of video recording applications in healthcare but in practice these have largely been largely confined to research, education, and quality improvement. Researchers value the richness of video data that includes sound, environmental context, body language and facial expressions, thus facilitating objective, accurate documentation of behaviour. In medical education, video-recordings assist clinicians in recognising visual and auditory clues during clinical consultations that cannot be derived from text-based learning. Video-based surgical records have informed quality improvement initiatives through the provision of increased detail and nuance beyond what exists in written operative notes alone. A further clear advantage of video recording is the creation of a permanent visual patient record that can be reviewed repeatedly by multiple professionals, ultimately increasing the accuracy of clinical assessment and improving communication among multi-professional healthcare workers.

Nevertheless, ethico-legal concerns and patient confidentiality have historically limited the use of video-recording for direct care purposes. Early studies suggested that patients can feel censored or self-conscious in front of a camera and video recording can have a detrimental impact on the therapeutic relationship. However, over the last decade, the proliferation of smartphones had led to video recordings being captured in everyday life, and technological advances are supporting lawful collection, handling, and storage of visual data to protect people's privacy in line with data protection legislation.

Little is known about how video recordings can support the safety and quality of individual patient care. Members of the study team recently conducted a systematic review to explore use of video-recording patients for direct care purposes. Twenty-seven studies published in the last 10 years were identified, evaluating acceptability, effectiveness, and/or ethico-legal considerations associated with video-recording patients to support care delivery. The review also brought together key guidance and recommendations of professional and regulatory bodies in the UK relating to audio-visual recording in healthcare. Evidence suggests that video recording patients for direct care purposes may be acceptable to patients and professionals, providing that the benefits are clear and risks are properly mitigated. Video technologies have been piloted in a variety of different health and care contexts to support diagnosis, care, and treatment, however, no studies have examined the application of video-based patient records for supporting older people's care transitions. Furthermore, the extent to which video recording is effective in support direct patient care remains unclear due the small number of published studies and poor quality of existing evidence.

Video recordings could enhance the safety and quality of care transitions for older people with frailty through providing objective and richly detailed visual information about their functional capabilities, support needs, and care preferences. However, making and sharing patient video recordings raises important ethical and legal considerations that must be addressed to enable the practical application of video for direct care purposes. This study will explore the acceptability, feasibility, and potential effectiveness of embedding in the electronic patient record, video recordings captured during routine care.

A programme theory (below), developed by our multidisciplinary steering group and informed by national frailty policy, suggests how video-based patient records could lead to patient benefit.

Programme Theory

If (1) it were acceptable and feasible to video-record frail, older patients, capturing their functional abilities, support needs, and care preferences at key timepoints (e.g. hospital discharge), and (2) the video-recordings were available for view by all those assessing/caring for the person across primary/secondary/community settings,

Then (3) A shared understanding of the person's functional abilities and support needs could be created, (4) A longitudinal view of the patient's function could be visualised, (5) Communication during patient handovers/at care interfaces could be improved,

So that (6) Older people with frailty receive care that is more person-centred and joined up, (7) Deterioration of frailty status is recognised and act upon earlier, (8) Improvements in care delivery can be achieved in line with the NHS Long Term Plan and the NHS RightCare Frailty Toolkit

So that (9) Older people with frailty suffer less avoidable complications and spend less time in hospital when they don't need to be there, and (10) Older people's experiences of care and health outcomes can be improved.

ELIGIBILITY:
Patients.

Inclusion Criteria:

* Admitted as an inpatient to an acute Medicine for the Elderly ward at St Mary's Hospital during a 3-month pilot phase of Isla's visual record platform
* Aged ≥65 years old
* Are considered to be frail or pre-frail by the direct care team
* Have capacity to consent to study participation OR lack capacity to consent on the condition that a 'personal consultee' is available to advise on the patient's likely wishes and feelings about taking part.

Exclusion Criteria:

* Patients who lack capacity to consent will be excluded if a personal consultee is not available to advise on the patients' likely wishes or feelings about taking part.

Carers.

Inclusion Criteria:

* Aged ≥18 years
* Provide the patient/care-recipient with assistance in their daily activities and are unpaid for these caring activities
* Are willing to participate in an interview as part of the study
* A carer may be a member of the patient's family, a friend, or other person who provides the patient with unpaid care

Exclusion Criteria:

- Carers will be excluded if the patient/care-recipient declined to participate in the study

Ward team.

Inclusion Criteria:

* Clinical staff working on an acute Medicine for the Elderly ward at St Mary's Hospital.
* Staff must be working regular shifts on the ward during study initiation and pilot phases
* Staff must have an active nhs.net account.

Exclusion Criteria:

* Ad-hoc bank/agency staff
* Permanent staff on long-term leave (e.g. sick/maternity) during the pilot

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients: Adults, aged 65 years or older, who are frail or pre-frail, and who are admitted as an inpatient to an acute Medicine for the Elderly ward during a three-month pilot phase
  Carers: Carers of enrolled patients, who provide the enrolled patient with assistance in their daily activities and are unpaid for these caring activities. A carer may be a member of the patient's family, a friend, or other person who provides the patient with unpaid care
  Ward team: Clinical staff working on one of three Medicine for the Elderly wards at St Mary's Hospital, where the Isla for Frailty intervention (described above) will be subject to a feasibility trial
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Intervention acceptability [1] | Within three-month pilot phase
  Patient and carer perspectives on the acceptability of video-based records will be assessed within this mixed-methods feasibility study and process evaluation multiple measures:
  [a] Proportion of eligible participants declining enrolment and reasons for non-participation (% declining, descriptive statistics)
Intervention acceptability [2] | Within three-month pilot phase
  Patient perspectives on the acceptability of video-based records will be assessed within this mixed-methods feasibility study and process evaluation multiple measures:
  [b] Proportion of enrolled patients with ≥ 1 video linked to the electronic patient record (% with at least one video linked to electronic patient record, descriptive statistics)
Intervention acceptability [3] | At or within two weeks of patient discharge
  Patient and carer perspectives on the acceptability of video-based records will be assessed within this mixed-methods feasibility study and process evaluation multiple measures:
  [c] Semi-structured interview at or within 2 weeks of discharge (Framework analysis to understand patient and carer views on acceptability)
Intervention acceptability [4] | Within three-month pilot phase
  Ward team perspectives on the acceptability of video-based records will be assessed within this mixed-methods feasibility study and process evaluation multiple measures:
  [a] Video evaluation questionnaire (a combination of stuctured and open-ended questions asking ward team to appraise whether video quality is suitable for clinical interpretation: Yes/No/To some extent; Video length: Too long/Too short/Just right, Whether ward team want to see more patient videos in the future: Yes/No - descriptive statistics. Open-ended questions ask ward team to explain their answers)
Intervention acceptability [5] | Ward staff interviews to be conducted within two months after three-month pilot phase
  Ward team perspectives on the acceptability of video-based records will be assessed within this mixed-methods feasibility study and process evaluation multiple measures:
  [b] Semi-structured interview after the three-month pilot (Framework analysis to understand ward team views on acceptability)
Intervention acceptability [6] | Within three-month pilot phase
  Ward team perspectives on the acceptability of video-based records will be assessed within this mixed-methods feasibility study and process evaluation multiple measures:
  [c] Number of videos requested, attempted & submitted (Quantitative, descriptive statistics)

SECONDARY OUTCOMES:
Intervention feasibility - Patient enrolment [1] | Within three-month pilot phase
  The feasibility of implementing a visual medical record platform (Isla) in the acute Medicine for the Elderly setting will be assessed within this mixed-methods feasibility study and process evaluation using multiple measures:
  [a] Proportion of eligible participants who were enrolled into the study (% enrolling, descriptive statistics)
Intervention feasibility - Patient enrolment [2] | Within three-month pilot phase
  The feasibility of implementing a visual medical record platform (Isla) in the acute Medicine for the Elderly setting will be assessed within this mixed-methods feasibility study and process evaluation using multiple measures:
  [b] Diversity of patient sample (Descriptive statistics to summarise sex; age; ethnicity; language spoken at home; Clinical Frailty Score [1-9]; dementia diagnosis [yes/no]; capacity to consent to study participation [yes/no] of patients who were enrolled, versus patients who declined participation)
Intervention feasibility - Intervention barriers and facilitators [1] | At or within two weeks of patient discharge
  The feasibility of implementing a visual medical record platform (Isla) in the acute Medicine for the Elderly setting will be assessed within this mixed-methods feasibility study and process evaluation using multiple measures:
  [a] Semi-structured interviews with patients/carers (Framework analysis to understand patient and carer views on intervention barriers and facilitators)
Intervention feasibility - Intervention barriers and facilitators [2] | Ward staff interviews to be conducted within two months after three-month pilot phase
  The feasibility of implementing a visual medical record platform (Isla) in the acute Medicine for the Elderly setting will be assessed within this mixed-methods feasibility study and process evaluation using multiple measures:
  [b] Semi-structured interviews with direct care team (Framework analysis to understand ward team views on intervention barriers and facilitators)
Intervention feasibility - Use of the Isla platform [1] | Within three-month pilot phase
  The feasibility of implementing a visual medical record platform (Isla) in the acute Medicine for the Elderly setting will be assessed within this mixed-methods feasibility study and process evaluation using multiple measures:
  [a] Proportion of enrolled patients with videos linked to the electronic patient record (% of patients with videos linked to electronic patient record, descriptive statistics)
Intervention feasibility - Use of the Isla platform [2] | Within three-month pilot phase
  The feasibility of implementing a visual medical record platform (Isla) in the acute Medicine for the Elderly setting will be assessed within this mixed-methods feasibility study and process evaluation using multiple measures:
  [b] Video view metrics (number of video views, descriptive statistics)
Intervention feasibility - Privacy and security concerns [1] | Within three-month pilot phase
  The feasibility of implementing a visual medical record platform (Isla) in the acute Medicine for the Elderly setting will be assessed within this mixed-methods feasibility study and process evaluation using multiple measures:
  [a] Number of videos raising cause for concern reported to the clinical lead (number of videos reported to clinical lead, descriptive statistics)
Perceived effectiveness of intervention [1] | Within three-month pilot phase
  The perceived effectiveness of patient videos for supporting elderly inpatient care (e.g. perceived impacts on inpatient assessment & clinical decision-making, multi-disciplinary team communication, care continuity during a hospital stay, person-centred care during a hospital stay) will be assessed within this mixed-methods feasibility study and process evaluation using multiple measures:
  [a] Video evaluation questionnaires (a combination of stuctured and open-ended questions asking ward team to appraise video usefulness for supporting patient assessment: Very useful/Somewhat useful/Useless; Usefulness of video for supporting decision-making: Very useful/Somewhat useful/Useless; Usefulness of video for communicating patient information to colleagues: Very useful/Somewhat useful/Useless - descriptive statistics. Open-ended questions ask ward team to explain their answers)
Perceived effectiveness of intervention [2] | Ward staff interviews to be conducted within two months after three-month pilot phase
  The perceived effectiveness of patient videos for supporting elderly inpatient care (e.g. perceived impacts on inpatient assessment & clinical decision-making, multi-disciplinary team communication, care continuity during a hospital stay, person-centred care during a hospital stay) will be assessed within this mixed-methods feasibility study and process evaluation using multiple measures:
  [b] Semi-structured interviews with direct care team after the pilot (Framework analysis to understand ward team views on perceived effectiveness)
Perceived effectiveness of [3] | At or within two weeks of patient discharge
  The perceived effectiveness of patient videos for supporting elderly inpatient care (e.g. perceived impacts on inpatient assessment & clinical decision-making, multi-disciplinary team communication, care continuity during a hospital stay, person-centred care during a hospital stay) will be assessed within this mixed-methods feasibility study and process evaluation using multiple measures:
  [c] Semi-structured interviews with patients/patient-carer dyads at or within 2 weeks of discharge (Framework analysis to understand patient and carer views on perceived effectiveness)

CONTACTS AND LOCATIONS:
Overall Officials: Phoebe Averill, PhD, Principal Investigator — Imperial College London
Locations (1):
- St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT06504641/Prot_000.pdf